CLINICAL TRIAL: NCT02445599
Title: Diclofenac Premedication, as the Effect of Preemptive Analgesia After Post-thoracotomy Chest and Shoulder Pain, as Well as the Changes of the Postoperative Breathing Function Values, a Randomized, Controlled, Prospective Trial
Brief Title: Diclofenac Premedication, as the Effect of Preemptive Analgesia After Post-thoracotomy Chest and Shoulder Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Debrecen (Other)
Responsible Party: Principal Investigator, Tamas Vegh, MD, MD, PhD assistant professor anesthesiologist and intensive care specialist, University of Debrecen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DEOEC RKEB/IKEB 4044-2013
Record Dates: First submitted 2014-12-11; First posted 2015-05-15 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Pain; Inadequate or Impaired Respiratory Function
Keywords: thoracotomy; pain management; analgesia; postoperative care; premedication; preventive
MeSH Terms: conditions — Pain; Respiratory Insufficiency; Agnosia | interventions — Diclofenac; Midazolam; Atropine; bucain; Fentanyl; Nalbuphine; Neodolpasse; Dipyrone; Tramadol

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diclofenac group (Experimental): Diclofenac 100 mg tablet were administered orally and Midazolam 5 mg + Atropine 0.5 mg were administered intramuscularly as premedication, 60 minutes before surgical interventions.
  Every patient recieved additional thoracic epidural analgesia during and after the surgery.
  As rescue medication patients get nalbuphine 10-20mg, diclofenac 75 mg + orphenadrine 30 mg (NEODOLPASSE infusion), metamizole-sodium 2g, tramadol 50-100mg as needed postoperatively.
  Interventions: Drug: Diclofenac; Drug: Midazolam; Drug: Atropine; Drug: bucain + fentanyl; Drug: Nalbuphine; Drug: Metamizole-sodium; Drug: Tramadol
- Control group (Experimental): Midazolam 5 mg + Atropine 0.5 mg were administered intramuscularly as premedication 60 minutes before surgical interventions.
  Every patient recieved additional thoracic epidural analgesia during and after the surgery.
  As rescue medication patients get nalbuphine 10-20mg, diclofenac 75 mg + orphenadrine 30 mg (NEODOLPASSE infusion), metamizole-sodium 2g, tramadol 50-100mg as needed postoperatively.
  Interventions: Drug: Midazolam; Drug: Atropine; Drug: bucain + fentanyl; Drug: Nalbuphine; Drug: Diclofenac; Drug: Metamizole-sodium; Drug: Tramadol

INTERVENTIONS:
Drug: Diclofenac — Orally 100 mg Diclofenac, administered 1 hour before surgery
  Other Names: Diclofenac Stada 100 mg retard
  Arms: Diclofenac group
Drug: Midazolam — 5 mg Dormicum intramuscularly, administered 1 hour before surgery
  Other Names: Dormicum 5mg/ml
Drug: Atropine — 0.5 mg Atropine intramuscularly, administered 1 hour before surgery
  Other Names: Atropine 1 mg/ml
Drug: bucain + fentanyl — Via the thocacic epidural cannula 1mg/ml bucain + 5microgr/ml fentanyl solution, with 0.1ml/kg body mass/hour speed is administered.
Drug: Nalbuphine — 1st choice for rescue analgetic 10-20 mg intravenously
  Other Names: Nubain 20mg/2ml
Drug: Diclofenac — 2nd choice for rescue analgetic 250ml intravenously
  Other Names: Neodolpasse 75 mg/ 250ml
Drug: Metamizole-sodium — Additional rescue analgetic 2g intravenously
  Other Names: Algopyrin 2g/2ml
Drug: Tramadol — Additional rescue analgetic 100mg intravenously
  Other Names: Contramal 100mg/2ml

SUMMARY:
The purpose of the study is to examine if the hyposthesis of the preventive analgestic characteristic of diclofenac given preoperatively has any effect on postoperative thoracic wall and shoulder pain sensation. We also want to examine the rescue analgetic consumption and the postoperative lung function test values.

DETAILED DESCRIPTION:
Introduction Thoracotomies are thought to be one of the most difficult surgical incisions to deal with post-operatively, because they are extremely painful and the pain can prevent the patient from breathing effectively. Currently in our institute the surgical and post-operative anelgesia are managed by the combination of local anesthetics and opioid pain killers through an epidural cannula. In addition the investigators give diclofenac intravenously (from the 2nd day after the operation per os) as well as nalbuphin is given intravenously to the patients if it is necesserary.

By definition pre-emptive analgesia means that the treatment of pain is initiated before the surgical procedure by analgetics or nerve blockade techniques. The purpose of this method is to inhibit the production of inflammatory mediators and the prevention of the pain stimulus entering the central nervous system. As a result of the pre-emptive antinociceptive treatment, the quantity of post-operative medications can be decreased, the analgesia has less complications and the patients are more satisfied.

In the study the researchers would like to examine the pre-emptive analgetic effect of diclofenac.

Patients and methods:

Patients undergoing thoracotomy are divided into two groups.:

* Study Group: 100mg diclofenac per os (n=50)
* Control Group: patients do not get diclofenac premedication (n=50) The investigators examine every patient for five days: they record the patients' pain with the help of the Visual Analogue Scale (VAS). We measure the analgetic consumption in intramuscular morphin equivalent dose and the local anesthetic consumption via epidural cannula seperately. The lung function testing was carried out two times postoperatively with the help of the MIR Spirolab II mobil spirometer.

ELIGIBILITY:
Inclusion Criteria:

* 100 thoracotomy patients who agreed to take part in our study and signed a consent
* age 18-80 years
* ASA I-III
* men/women equally
* thoracotomies are managed with using intratracheal double lumen tube
* insertion of thoracic epidural cannula and during the operation administration of 1mg/ml bucain, 5microgr/ml fentanyl solution, with 0.1ml/kg body mass/hour speed

Exclusion Criteria:

* acute operation
* diclofenac allergy in the anamnesis
* the lack of thoracic epidural cannula

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
10% reduction of the thoracotomy pain recorded by VAS score. | 5 days
  Our main goal is to achieve 10% reduction of the thoracotomy pain recorded by VAS score, compared to the non-diclofenac control group.

SECONDARY OUTCOMES:
10% reduction of the shoulder pain recorded by VAS score. | 5 days
  Our second goal is to achieve 10%reduction of the shoulder pain recorded by VAS score, compared to the non-diclofenac control group.

OTHER OUTCOMES:
Analgetic need during the first five postoperative days. | Participants were followed for 5 days postoperatively
  The total amount of administered analgetics were recorded during the first five postoperative days and then converted into intramuscular morphine equivalents.
Postoperative complications during the first five postoperative days | Participants were followed for 5 days postoperatively
  Intraoperative fentanyl use was registered as micrograms per kilogram body weight and micrograms per hour as well.
  Postoperative complications such as bleeding at the surgical site, gastrointestinal problems or kidney dysfunctions were also registered.
Intraoperative fentanyl use | Participants were followed during the operation on day 1
  Intraoperative fentanyl use was registered as micrograms per kilogram body weight and micrograms per hour as well.
Epidurally administered local anethetics | Participants were followed for 5 days postoperatively
  The total amount of epidurally administered local anesthetic were recorded during the first five postoperative days.
Comparing the pre- and postoperative lung function test values | Participants were followed for 5 days postoperatively
  Comparing the pre- and postoperative lung function test values with and after the removal of chest drains. The measurement were executed by the MIR Spirolab II bedside spirometer.

CONTACTS AND LOCATIONS:
Overall Officials: Béla Fülesdi, MD,PhD,DSci, Principal Investigator — UNIVERSITY OF DEBRECEN FACULTY OF MEDICINE Department of Anesthesiology and Intensive Care Debrecen, Hungary, 4032
Locations (1):
- UNIVERSITY OF DEBRECEN FACULTY OF MEDICINE Department of Anesthesiology and Intensive Care, Debrecen, Hajdú-Bihar, Hungary

REFERENCES:
- [Background] Gerner P. Postthoracotomy pain management problems. Anesthesiol Clin. 2008 Jun;26(2):355-67, vii. doi: 10.1016/j.anclin.2008.01.007. PMID 18456219
- [Background] Gottschalk A, Cohen SP, Yang S, Ochroch EA. Preventing and treating pain after thoracic surgery. Anesthesiology. 2006 Mar;104(3):594-600. doi: 10.1097/00000542-200603000-00027. No abstract available. PMID 16508407
- [Background] Koehler RP, Keenan RJ. Management of postthoracotomy pain: acute and chronic. Thorac Surg Clin. 2006 Aug;16(3):287-97. doi: 10.1016/j.thorsurg.2006.05.006. PMID 17004557
- [Background] Ochroch EA, Gottschalk A. Impact of acute pain and its management for thoracic surgical patients. Thorac Surg Clin. 2005 Feb;15(1):105-21. doi: 10.1016/j.thorsurg.2004.08.004. PMID 15707349
- [Background] McCormack HM, Horne DJ, Sheather S. Clinical applications of visual analogue scales: a critical review. Psychol Med. 1988 Nov;18(4):1007-19. doi: 10.1017/s0033291700009934. PMID 3078045
- [Background] Gotoda Y, Kambara N, Sakai T, Kishi Y, Kodama K, Koyama T. The morbidity, time course and predictive factors for persistent post-thoracotomy pain. Eur J Pain. 2001;5(1):89-96. doi: 10.1053/eujp.2001.0225. PMID 11394926
- [Result] Nesek-Adam V, Grizelj-Stojcic E, Mrsic V, Rasic Z, Schwarz D. Preemptive use of diclofenac in combination with ketamine in patients undergoing laparoscopic cholecystectomy: a randomized, double-blind, placebo-controlled study. Surg Laparosc Endosc Percutan Tech. 2012 Jun;22(3):232-8. doi: 10.1097/SLE.0b013e31824f8ae4. PMID 22678319